CLINICAL TRIAL: NCT02183298
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Doses (0.5 mg to 10 mg) of BI 1356 BS as Formulation for Intravenous Administration in Healthy Male Volunteers. A Randomised, Single-blind, Placebo-controlled Trial, Including a Crossover Intra-subject Bioavailability Comparison of 5 mg BI 1356 BS iv Solution and 10 mg BI 1356 BS as Tablet.
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Doses of BI 1356 BS in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1218.10
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin

ARMS (2):
- BI 1356 BS - single rising dose (Experimental)
  Interventions: Drug: BI 1356 BS - intravenous; Drug: BI 1356 BS - Tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1356 BS - intravenous
  Arms: BI 1356 BS - single rising dose
Drug: BI 1356 BS - Tablet
  Arms: BI 1356 BS - single rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of BI 1356 as formulation for intravenous administration

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests
* Age ≥18 and Age ≤50 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsade de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Exclusion criteria specific for this study:

* Veins unsuitable for infusion
* PR interval >220 ms or QRS interval >120 ms

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Screening, up to 14 days following drug administration
Number of patients with clinically changes in vital signs (blood pressure [BP], pulse rate [PR]) | Screening, up to 14 days following drug administration
Number of patients with abnormal findings in 12-lead ECG (electrocardiogram) | Screening, up to 14 days following drug administration
Number of patients with abnormal changes in laboratory parameters | Screening, up to 14 days following drug administration
Number of patients with adverse events | up to 35 days
Assessment of tolerability by investigator on a 4-point scale | up to 14 days following drug administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | predose, up to 192 h following drug administration
tmax (time from dosing to maximum measured concentration) | predose, up to 192 h following drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | predose, up to 192 h following drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | predose, up to 192 h following drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | predose, up to 192 h following drug administration
λz (terminal rate constant in plasma) | predose, up to 192 h following drug administration
t1/2 (terminal half-life of the analyte in plasma) | predose, up to 192 h following drug administration
MRT/ MRTpo (mean residence time of the analyte in the body after iv/oral administration) | predose, up to 192 h following drug administration
CL/ CL/F (total clearance of the analyte in plasma after iv/oral administration) | predose, up to 192 h following drug administration
Vz/ Vz/F (apparent volume of distribution during the terminal phase λz following an iv/oral dose) | predose, up to 192 h following drug administration
Vss (apparent volume of distribution at steady state following intravascular administration) | predose, up to 192 h following drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | predose, up to 120 h following drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | predose, up to 120 h following drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | predose, up to 120 h following drug administration
Changes of Dipeptidyl-Peptidase IV (DPP-IV) activity in plasma | up to 192 h following drug administration